CLINICAL TRIAL: NCT03887299
Title: Antimicrobial Dressing Versus Standard Dressing in Obese Women Undergoing Cesarean Delivery: A Randomized Control Trial
Brief Title: Antimicrobial Dressing Versus Standard Dressing in Obese Women Undergoing Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-0265
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2019-03

CONDITIONS: Cesarean Section Complications; Wound Breakdown; Wound Infection; Satisfaction; Surgical Wound Infection
Keywords: Cesarean; Wound care; Wound complication; Surgical site infection
MeSH Terms: conditions — Surgical Wound Dehiscence; Wound Infection; Personal Satisfaction; Surgical Wound Infection | interventions — Chromogranins

STUDY DESIGN:
Intervention Model Description: Open label randomized control trial
Masking Description: Data analysis will be blinded to assignment including the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Wound Care (Placebo Comparator): Wound dressing and care as per our current practice. Compression dressing consisting of gauze, tefla and adhesive tape will be placed intraoperatively. Dressing will be removed after 24 hours from surgery completion and subjects will have an absorption pad with overlying garments for the remaining postoperative days until standard postoperative visit for wound check.
  Interventions: Other: Standard Wound Care
- CHG Wound Care (Active Comparator): ReliaTect™ Post-Op Dressing will be applied as per the manufacturer's instructions intraoperatively. The dressing will be in place until the postoperative clinic visit on postoperative day 7.
  Interventions: Combination Product: ReliaTect™ Post-Op Dressing (contains chlorohexidine gluconate or CHG)

INTERVENTIONS:
Combination Product: ReliaTect™ Post-Op Dressing (contains chlorohexidine gluconate or CHG) — Dressing will be applied in the operating room at the end of case and be in place until postoperative day 7
  Other Names: Dressing containing CHG a disinfectant and antiseptic that is used for skin disinfection
  Arms: CHG Wound Care
Other: Standard Wound Care — Wound care will be administered as standard protocol in our institution
  Arms: Standard Wound Care

SUMMARY:
This will be an open label pilot randomized controlled clinical trial. Women undergoing cesarean delivery will be randomized to have standard wound dressing care or chlorohexidine gluconate (CHG) impregnated wound dressing (ReliaTect™ Post-Op Dressing).

DETAILED DESCRIPTION:
Subjects requiring cesarean delivery and without exclusion criteria will be informed by the obstetrical team about the study and asked for permission to contact the study personnel. Written informed consent will be obtained by person-to-person contact. The research staff will be responsible for the informed consent.

Subjects who agree to participate in the study will be randomized to one of the two groups below in a 1/1 allocation:

* Standard Wound Care: Wound dressing and care as per our current practice. Compression dressing consisting of gauze, tefla and adhesive tape will be placed intraoperatively. Dressing will be removed after 24 hours from surgery completion and subjects will have an absorption pad with overlying garments for the remaining postoperative days until standard postoperative visit for wound check.
* CHG Wound Care: ReliaTect™ Post-Op Dressing will be applied as per the manufacturer's instructions (Appendix A) intraoperatively. The dressing will be in place until the postoperative clinic visit on postoperative day 7.

The remainder of the subjects' care will be similar for both arms and will follow current standard clinical practice at the University of Texas Medical Branch (UTMB).

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age.
* Women ≥ 24 weeks' viable gestation.
* To undergo cesarean delivery.
* Admission BMI ≥ 35.

Exclusion Criteria:

* Patient unwilling or unable to provide consent.
* No prenatal care or a non-resident patient who is unlikely to be followed-up after delivery.
* Immunosuppressed subjects: i.e., taking systemic immunosuppressant or steroids (e.g. transplant subjects; not including steroids for lung maturity), HIV with CD4 <200, or other.
* Decision not to have skin closure (e.g. secondary wound closure, mesh closure).
* Current skin infection.
* Coagulopathy.
* High likelihood of additional surgical procedure beyond cesarean (e.g. scheduled hysterectomy, bowel or adnexal surgery).
* Known allergy to CHG.
* Incarcerated individuals.
* Chorioamnionitis.
* Subjects participating on other treatment trials or studies that would interfere with the current study's primary outcome.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Obstetrical population: Pregnant women undergoing cesarean section
Enrollment: 154 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio F. Saad, MD, Principal Investigator — UTMB Galveston
Locations (1):
- Ashley Salazar, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allegranzi B, Zayed B, Bischoff P, Kubilay NZ, de Jonge S, de Vries F, Gomes SM, Gans S, Wallert ED, Wu X, Abbas M, Boermeester MA, Dellinger EP, Egger M, Gastmeier P, Guirao X, Ren J, Pittet D, Solomkin JS; WHO Guidelines Development Group. New WHO recommendations on intraoperative and postoperative measures for surgical site infection prevention: an evidence-based global perspective. Lancet Infect Dis. 2016 Dec;16(12):e288-e303. doi: 10.1016/S1473-3099(16)30402-9. Epub 2016 Nov 2. PMID 27816414
- [Background] Berg CJ, Chang J, Callaghan WM, Whitehead SJ. Pregnancy-related mortality in the United States, 1991-1997. Obstet Gynecol. 2003 Feb;101(2):289-96. doi: 10.1016/s0029-7844(02)02587-5. PMID 12576252
- [Background] DeFrances CJ, Cullen KA, Kozak LJ. National Hospital Discharge Survey: 2005 annual summary with detailed diagnosis and procedure data. Vital Health Stat 13. 2007 Dec;(165):1-209. PMID 18350768
- [Background] Gibbs RS. Clinical risk factors for puerperal infection. Obstet Gynecol. 1980 May;55(5 Suppl):178S-184S. doi: 10.1097/00006250-198003001-00045. PMID 6990333
- [Derived] Saad AF, Salazar AE, Allen L, Saade GR. Antimicrobial Dressing versus Standard Dressing in Obese Women Undergoing Cesarean Delivery: A Randomized Controlled Trial. Am J Perinatol. 2022 Jul;39(9):951-958. doi: 10.1055/s-0040-1721112. Epub 2020 Dec 2. PMID 33264808

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Wound Care | CHG Wound Care
Started | 77 | 77
Completed | 77 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Wound Care | CHG Wound Care | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Continuous [Median (Full Range); unit: years] | 29 [20 to 41] | 29 [19 to 41] | 29 [19 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 77 | 154
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 47 | 84
  Not Hispanic or Latino | 40 | 30 | 70
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 77 | 77 | 154
Medical Condition [Count of Participants; unit: Participants] | 27 | 23 | 50
Delivery complications [Count of Participants; unit: Participants] | 12 | 8 | 20
Vertical Skin incision [Count of Participants; unit: Participants] | 8 | 6 | 14
Skin closure with staples [Count of Participants; unit: Participants] | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction and QoL Questionnaire
Description: We will be assessing through a survey patient satisfaction concerning dressing received and assess the quality of life while receiving either intervention (5 point Richter scale). A maximum score of 5: Strongly agree and a minimum score of 1: Strongly disagree.
  A higher score means a better outcome.
Time Frame: Postpartum wound care visit (up to 10days postpartum)
Measure: Median (Full Range); unit: Score
Arm/Group | Standard Wound Care | CHG Wound Care
Number analyzed (Participants) | 77 | 77
Score | 49 [20 to 55] | 52 [12 to 55]

2. Secondary Outcome: Number of Participants With Composite Wound Complication
Description: Defined as presence of any of the following within 30 days from surgery: Wound infection: Presence of either superficial or deep incisional SSI described as cellulitis/erythema and induration around the incision or purulent discharge from the incision site, with or without fever, such as necrotizing fasciitis (diagnosed based on necrotizing wound infection). Wound hematoma, seroma, or breakdown alone. (yes or No)
Time Frame: 30 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Wound Care | CHG Wound Care
Number analyzed (Participants) | 77 | 77
Participants | 5 | 9

3. Secondary Outcome: Number of Participants With Wound Breakdown
Description: Opening of wound incision documented in the chart at the provider's discretion(Yes or No)
Time Frame: 30 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Wound Care | CHG Wound Care
Number analyzed (Participants) | 77 | 77
Participants | 1 | 0

4. Secondary Outcome: Number of Participants That Resulted in Maternal Death
Description: Death of participant during hospital stay (Yes or No)
Time Frame: 4 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Wound Care | CHG Wound Care
Number analyzed (Participants) | 77 | 77
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Puerperal Fever
Description: Temperature > 100.4oF after first 24 hours or ≥101 oF any time. (Yes or No)
Time Frame: 4 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Wound Care | CHG Wound Care
Number analyzed (Participants) | 77 | 77
Participants | 0 | 1

6. Secondary Outcome: Provider Satisfaction
Description: Assessing health care providers opinion on the dressing care (5 point Richter scale). A maximum score of 5: Strongly agree and a minimum score of 1: Strongly disagree.
  A higher score means a better outcome.
Time Frame: Postpartum wound care visit (up to 10days postpartum)
Measure: Median (Full Range); unit: Score
Arm/Group | Standard Wound Care | CHG Wound Care
Number analyzed (Participants) | 77 | 77
Score | 17 [5 to 25] | 21 [5 to 25]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 9 months from subject randomization.
Arm/Group | Standard Wound Care | CHG Wound Care
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT03887299/Prot_SAP_001.pdf